CLINICAL TRIAL: NCT03790501
Title: Impact of Physical Activity Routines and Dietary Intake on the Longitudinal Symptom Experience of People Living With HIV
Brief Title: Impact of Physical Activity and Diet on Symptom Experience in People Living With HIV
Acronym: PROSPER-HIV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: University of Alabama at Birmingham (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Allison Webel, Assistant Professor, University of Washington
Other Study IDs: STUDY00013048; R01NR018391 (NIH)
Record Dates: First submitted 2018-12-28; First posted 2018-12-31 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People living with HIV (PLHIV).: We will recruit and enroll 850 people living with HIV (PLHIV) to participate in this longitudinal observational study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — As an observational study, no intervention will be associated with the study group.

SUMMARY:
We will conduct a four-year, observational study of 850 participants to measure physical activity and diet, once a year for three years. All participants will also complete the standard Centers for AIDS Research (CFAR) Network of Integrated Clinical Systems (CNICS) patient-reported outcomes (PRO) and clinical assessment procedures. An enhanced PRO assessment (consisting measures of physical activity, diet intake and anthropomorphic factors) will be included after the routine patient clinic visit at four CNICS sites: Case Western Reserve University, University of Alabama at Birmingham, University of Washington, and Fenway Health.

DETAILED DESCRIPTION:
PROSPER-HIV is a four-year, prospective, observational study of 850 CNICS participants who will complete an enhanced patient-reported outcome (PRO) assessment to measure physical activity and diet intake, once a year for three years. All participants will also complete the standard CNICS PRO and clinical assessment procedures. We propose to integrate the following measures, physical activity (triaxial accelerometery), dietary intake (24-hour diet recalls), and anthropomorphic factors (waist-hip-ratio), into an enhanced annual assessment of patient reported outcomes at four CNICS sites: Case Western Reserve University, University of Alabama at Birmingham, University of Washington, and Fenway Health. Our four primary objectives are to:

1. Identify and characterize longitudinal, objectively measured, physical activity and dietary patterns among PLHIV
2. Examine the relationship between objectively-measured physical activity and self-reported physical activity on the Lipid Research Clinics Physical Activity Questionnaire.
3. Determine which aspects of physical activity patterns and diet quality are associated with decreased symptom burden and intensity in PLHIV, and if this relationship is moderated by age and sex.
4. Explore the potential mediating effect of anthropomorphic and physical fitness variables on the relationships between physical activity, dietary patterns, and symptom burden and intensity in PLHIV.

We hypothesize that people living with HIV who 1) have more intense, frequent and longer physical activity bouts will have age- and sex-dependent reduced symptom burden; 2) eat better quality diets (e.g., more fiber and protein, fewer carbohydrates) will have reduced symptom burden and intensity and that this relationship will also vary by age and sex.

ELIGIBILITY:
Inclusion Criteria:

1. Be an active CNICS participant
2. aged ≥18 years
3. prescribed HIV antiretroviral therapy, and
4. have an undetectable HIV viral load: defined as the most recent HIV viral load <200 copies/mL, checked within the past year.

Exclusion Criteria:

1) Did not complete the HIV Symptom Index in the PRO assessment (2) No reliable access to a telephone or internet-enable telephone services needed to complete the 24-diet recalls (3) Was pregnant, breast-feeding, or planning a pregnancy at the time of PRO assessment (4) Planning to move out of the area in the next 36 months, or (5) Non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit and enroll 850 people living with HIV (PLHIV) who participate in the Centers for AIDS Research Network of Integrated Clinical Systems cohort to participate in this longitudinal observational study.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Symptom Distress | Four years
  Symptom distress will be measured with the-20 item HIV Symptom Index. As recommended, our primary endpoints include 1) total symptom count (sum all symptoms that are reported as having the symptom and it bothers the participant at least a little); and 2) a total count of symptoms that bother the participant a lot (high symptom distress).

CONTACTS AND LOCATIONS:
Overall Officials: Allison Webel, BSN, PhD, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Fenway Institute, Boston, Massachusetts
  - Case Western Reserve University, Cleveland, Ohio
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared consistent with the CNICS Data Sharing Policy found here: https://www.uab.edu/cnics/images/CNICSdatasharing_policy_v081515.pdf
Supporting Information: Study Protocol, ICF
URL: https://www.uab.edu/cnics/images/CNICSdatasharing_policy_v081515.pdf

REFERENCES:
- [Derived] Horvat Davey C, Willig AL, Ruderman SA, Dos Santos AP, Oliveira V, Gripshover BM, Long DM, Cleveland JD, Crane HM, Fleming J, Buford TW, Burkholder G, Saag MS, Webel AR. Exploring the Relationship Between Insomnia and Biological Factors, Substance Use, and Physical Activity in People With HIV in the United States: Insights From the PROSPER Study. J Assoc Nurses AIDS Care. 2026 Jan-Feb 01;37(1):52-62. doi: 10.1097/JNC.0000000000000589. Epub 2025 Oct 1. PMID 41026762
- [Derived] Oliveira VHF, Willig AL, Horvat Davey C, Buford TW, Menezes P, Cachay E, Crane HM, Burkholder GA, Gripshover BM, Fleming JG, Cleveland JD, Webel AR. Brief Report: Relationship Between Adiposity and Biomarkers of Aging and Frailty Among Adults Aging With HIV. J Acquir Immune Defic Syndr. 2024 Apr 1;95(4):377-382. doi: 10.1097/QAI.0000000000003362. PMID 38100820
- [Derived] Webel AR, Davey CH, Oliveira V, Cleveland D, Crane HM, Gripshover BM, Long DM, Fleming JG, Buford TW, Willig AL. Physical activity is associated with adiposity in older adults with HIV in the modern HIV era. AIDS. 2023 Oct 1;37(12):1819-1826. doi: 10.1097/QAD.0000000000003635. Epub 2023 Jun 27. PMID 37382891
- [Derived] Webel AR, Long D, Rodriguez B, Davey CH, Buford TW, Crane HM, Mayer K, Saag MS, Willig AL. The PROSPER-HIV Study: A Research Protocol to Examine Relationships Among Physical Activity, Diet Intake, and Symptoms in Adults Living With HIV. J Assoc Nurses AIDS Care. 2020 May-Jun;31(3):346-352. doi: 10.1097/JNC.0000000000000145. No abstract available. PMID 31789686